CLINICAL TRIAL: NCT04537767
Title: The Effect of Esmolol on Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES-01
Record Dates: First submitted 2020-06-14; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Sepsis
Keywords: sepsis; septic shock; esmolol
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): Patients randomly assigned to the ES group were treated with esmolol to control the heart rate to the target range.
  Interventions: Drug: Esmolol
- control group (Placebo Comparator): Patients randomly assigned to the control group were treated with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmolol — The protocol required a titrated esmolol infusion commenced at 25 mg/ h, with an upper dose limit of 2000 mg/h, to maintain the HR between 75 and 90 bpm in ES group. The control group were treated with placebo.
  Arms: ES group
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
The investigators conduct an RCT to explore the efficacy of esmolol in patients with septic shock and sepsis.

DETAILED DESCRIPTION:
Severe sepsis, septic shock, and their complications have become the major healthcare problem that affects millions of people each year, resulting in high mortality rates. Septic responses have an extremely complex chain of events including inflammatory and anti-inflammatory processes, humoral and cellular reactions, and cardiocirculatory abnormalities. Esmolol may have some potential in treating septic shock and sepsis. The investigators conduct an RCT to explore the efficacy of esmolol in patients with septic shock and sepsis.

ELIGIBILITY:
Inclusion Criteria:

* sepsis patients
* HR>100bpm 6h after admission
* with CVC and ScvO2>65%

Exclusion Criteria:

* age <18 years,
* used β-blocker before,
* cardiac dysrhythmias,
* need for an inotropic agent,
* valvular heart disease,
* hemoglobin>6g/L
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
REE | Day 7 after enrollment
  Resting energy expenditure

SECONDARY OUTCOMES:
28-day mortality rate | Day 28 after enrollment
  28-day mortality rate
HR control rate | 24 hours after enrollment
  target heart rate control rate
Vasoactive drug administration dose | Day 1/3/7 after enrollment
  Vasoactive drug administration dose
Concentration of Lac | Day 1/3/7 after enrollment
  Concentration of lactic acid
O2ER | Day 1/3/7 after enrollment
  oxygen extraction rate

IPD SHARING:
Plan to Share IPD: No